CLINICAL TRIAL: NCT05107609
Title: Psychobiological Processes in Social Evaluation: Pilot Testing a Self-Compassion Intervention for Weight Stigma
Brief Title: Psychobiological Processes in Social Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Eva Pila, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-0000-E
Record Dates: First submitted 2021-08-20; First posted 2021-11-04 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Stigma, Social; Weight, Body; Compassion; Stress Reaction
MeSH Terms: conditions — Social Stigma; Body Weight; Fractures, Stress

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be aware that they are randomized into one of two intervention conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention (Experimental): Participants will be guided through an acute, 30-minute self-compassion intervention consisting of psychoeducation, guided loving-kindness meditation, compassionate imagery and a compassionate writing activity.
  Interventions: Behavioral: Acute Self-Compassion Intervention
- Resting Control Intervention (No Intervention): Participants will be asked to sit quietly and independently for 30 minutes. They can read neutral magazines provided or their own reading/writing material, but will be asked not to use outside electronic devices or communicate with anyone external.

INTERVENTIONS:
Behavioral: Acute Self-Compassion Intervention — Participants will be guided through a 30-minute behavioural self-compassion intervention that seeks to mitigate their psychobiological responses to the subsequent weight stigma induction. The intervention is intended to induce a flexible self-compassionate mindset that will facilitate more adaptive psychological responding to stress and activate affiliative/self-soothing physiological systems that can dampen psychobiological stress reactivity. This acute self-compassion intervention will employ a multimodal, experiential approach that is regularly utilized in self-compassion training, drawing from approaches developed in Compassion-Focused Therapy and Mindful Self-Compassion.
  Arms: Self-Compassion Intervention

SUMMARY:
Higher-weight individuals face pervasive weight-related stigma and discrimination in their daily lives. There is conceptual and empirical evidence to suggest that weight stigma contributes to worse physical and psychological health outcomes, mediated by the deleterious psychobiological responses to psychosocial stress. Activating self-soothing emotional states (such as self-compassion) may protect against this psychobiological cascade, conferring resilience to negative social evaluation (such as weight stigma). This proof-of-concept study aims to establish the feasibility of an experimental protocol testing whether an acute self-compassion intervention can attenuate the psychobiological stress response to induced weight-based social-evaluative threat. Participants will be randomized into either self-compassion intervention or rest control groups. A standard body composition assessment will be used to induce weight stigma among young women who self-identify as "higher-weight." Stress-sensitive biomarkers (i.e., salivary cortisol and heart-rate variability) along with psychological indices of self-conscious emotions will be used to quantify the psychobiological stress response. This novel pilot study will contribute to efforts to understand the psychobiological processes by which self-compassion facilitates adaptive responding to acute stress, and will help inform future tests of interventions focused on mitigating the harmful health effects of social stigma.

DETAILED DESCRIPTION:
This is a randomized proof-of-concept experiment with two conditions: self-compassion intervention and no-intervention (i.e., quiet rest) control.

The primary objective of this pilot study is to examine the feasibility and establish parameter estimates for a laboratory protocol to quantify the psychobiological responses to a lab-based weight stigma induction. Feasibility will include process assessments (i.e., examine acceptability of both the self-compassion intervention and weight stigma induction to participants, establish feasibility of recruitment goals and examine participant demand), resource assessment (i.e., test the practicality of the proposed experimental protocol), management assessment (i.e., test research group's ability to implement experimental protocol including self-compassion intervention, weight-based social-evaluative induction and biological biomarker collection), and scientific assessment (i.e., establish parameter estimates for psychological and biological responses to self-compassion intervention and social-evaluative threat induction). Due to the unpredictable nature of the COVID context for biological sample collection, no a prior criteria for feasibility are established.

The secondary objective is to perform limited-efficacy testing of the self-compassion intervention in reducing the psychobiological stress response relative to control condition. Efficacy will be assessed by comparing pre/post manipulation biological (i.e., cortisol, heart rate variability) and psychological (i.e., state shame, guilt, distress, internalized weight bias) indices between conditions (i.e., self-compassion intervention, rest control).

N=60 young adult cis-gender women who perceive themselves to be "heavier-weight" will be recruited to participate. After a brief telephone pre-screening interview to determine eligibility, participants will book two lab visits to complete a baseline assessment and experimental manipulation.

The first in-lab session will comprise of the informed consent process and computerized surveys to collect demographic and psychological baseline measures. This session will also serve as acclimatization to the lab environment, to minimize anticipatory anxiety and/or novel environment effects that may confound psychobiological stress measures during the experimental manipulation. After providing written informed consent, participants will complete a computerized survey consisting of demographic and baseline psychological measures.

All experimental sessions will take place between 1 pm and 5 pm to control for diurnal variation in cortisol and will be conducted in a light- and temperature-controlled laboratory. Participants will fill out a computerized survey to assess baseline psychological indices, and will provide a 5-minute baseline heart-rate variability measurement and saliva sample (#1).

Participants will be randomized into one of two experimental conditions: acute self-compassion intervention or rest control. Over the next 30 minutes, participants who were randomized into the self-compassion condition will be guided through a multi-modal behavioural self-compassion intervention. Participants in the no-intervention (resting) control group will be asked to sit quietly for 30 minutes. Immediately after the self-compassion induction (or control), participants will complete a measure of state self-compassion as a manipulation check and will repeat state psychological measures taken at baseline.

An anthropometric assessment including a standard three-site (triceps, iliac crest, thigh) skinfold body composition assessment, height and weight measurements will be performed by two thin researchers to induce weight stigma. Participants will undergo the assessment while wearing a physically revealing outfit (i.e., sports bra and spandex shorts) which they will be asked to change into at the beginning of the weight-stigma induction. This paradigm has been shown to successfully induce social evaluative threat in young women, eliciting cortisol and body shame responses.

Immediately after the weight stigma induction, participants will be asked to complete a brief survey assessing psychological outcome measures and to provide a saliva sample (#2). Then, participants will be asked to wait quietly for a 35-minute minute recovery phase, during which saliva samples will again be collected at 10 (#3), 20 (#4) and 35-minutes (#5) post-stressor.

After the recovery session is over, participants will be asked to respond to open-ended funnel debriefing questions to assess the believability of the cover story and the success of deception. Participants will also be asked questions related to the acceptability of the experimental protocol and social-evaluative induction. Finally, participants will be fully debriefed.

ELIGIBILITY:
Inclusion Criteria:

* Can read and communicate in English to provide informed consent
* Cis-gender woman (self-reports their gender as woman and assigned sex at birth as female)
* Age 18-34 inclusive
* Self-identify as "heavy weight"
* Currently taking oral contraceptives

Exclusion Criteria:

* Current smoking; current other nicotine/tobacco use; or current recreational drug use
* Current and active use of any oral prescription medication to treat a chronic health condition - excepting contraceptives
* Chronic health conditions as diagnosed by a licensed medical professional such as psychiatric (including substance use disorder, eating disorder), endocrine, cardiovascular, respiratory, autoimmune or other chronic conditions - excepting obesity, which will still be included due to inconsistent findings regarding whether obesity impacts neuroendocrine stress responses.
* Fever or acute illness/infection on day of experiment
* Pregnant or currently breastfeeding
* Prior experience with self-compassion training or compassion interventions, or prior experience with formal mindfulness or meditation training.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must identify as cis-gender women (i.e., self-report their gender identity as woman and self-report their assigned sex at birth as female)
Enrollment: 37 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Area under the curve for cortisol reactivity | Saliva samples will be collected at baseline, post-stigma induction (0 minutes), and at 10 (i.e. ~25 minutes post stressor onset, expected peak), 20 and 35 minutes post-induction
  Salivary cortisol will be used to quantify hypothalamic pituitary adrenal axis reactivity. Salivary cortisol concentration will be determined using a commercial high sensitivity EIA kit (Salimetrics; Carlsbad, CA). All assessments will be used to calculate area under the curve with respect to ground, and area under the curve with respect to increase.
Change in State Distress from baseline to post-stigma induction | Self-reported distress will measured at 3 points: baseline (~10 minutes after start of session), post self-compassion intervention or control (45 minutes after start) and post stigma induction (60 minutes after start).
  State distress will be measured using a modified version of widely-used single-item Subjective Units of Distress scale (SUDS; Wolpe, 1990) requiring participants to indicate their current distress level on a visual analog scale (VAS) of 1-100 (where 1 is low distress and 100 is high distress).
Change in State Self-Conscious Body Emotions from baseline to post-stigma induction | Self-report body emotions will measured at 3 points: baseline (~10 minutes after start of session), post self-compassion intervention or control (45 minutes after start) and post stigma induction (60 minutes after start).
  Purpose-built 4-item measure to assess the degree to which a participant feels self-conscious emotions about their body right now (i.e., body shame, body guilt, body embarrassment, body envy). Participants answer on a 5-point scale from 1 (very slightly or not at all) to 5 (extremely), where higher scores indicate greater levels of self-conscious body emotions.
Change in State Shame and Guilt from baseline to post-stigma induction | Self-report shame and guilt will measured at 3 points: baseline (~10 minutes after start of session), post self-compassion intervention or control (45 minutes after start) and post stigma induction (60 minutes after start)
  State Shame and Guilt Scale will quantify state shame and guilt. Participants indicate how each prompt describes how they are feeling right now on a 5-point scale: 1 = I do not feel this way at all; 3 = I feel this way somewhat; 5 = I feel this way very strongly. Higher scores indicate higher levels of state shame and guilt.
Change in State Weight Bias Internalization from baseline to post-stigma induction | Self-report weight bias internalization measured at 3 points: baseline (~10 minutes after session start), post self-compassion intervention or control (45 minutes after start) and post induction (60 minutes after start).
  Modified Weight Bias Internalization Scale will be modified to capture state-level weight bias internalization. Participants respond to each prompt on a 7-point scale from 1 (strongly disagree) to 7 (strongly agree), where higher scores indicate greater internalized weight bias.
Root mean square of successive differences in Heart Rate Variability (HRV) | 4 phases: baseline measurement (minutes 5-10), intervention (minutes 15-45), weight-stigma induction (minutes 45-60), recovery (minutes 60-95).]
  Data from all phases will be used to calculate root mean square of successive differences (RMSSD) will be used to quantify vagally-mediated HRV (i.e., parasympathetic cardiac activity).

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bargh, J. A., & Chartrand, T. L. (2000). The mind in the middle: A practical guide to priming and automaticity research. In H. T. Reis & C. M. Judd (Eds.), Handbook of research methods in social and personality psychology (pp. 253-285). Cambridge University Press.
- [Background] Cloudt MC, Lamarche L, Gammage KL. The impact of the amount of social evaluation on psychobiological responses to a body image threat. Body Image. 2014 Sep;11(4):350-6. doi: 10.1016/j.bodyim.2014.06.003. Epub 2014 Jun 28. PMID 24981013
- [Background] Jackson AS, Pollock ML, Ward A. Generalized equations for predicting body density of women. Med Sci Sports Exerc. 1980;12(3):175-81. PMID 7402053
- [Background] Lamarche, L., Gammage, K., Klentrou, P., Kerr, G., & Faulkner, G. (2014). Examining psychobiological responses to an anticipatory body image threat in women. Journal of Applied Biobehavioral Research, 19. doi: 10.1111/jabr.12022.
- [Background] Lamarche, L., Gammage, K. L., Kerr, G., Faulkner, G., & Klentrou, P. (2016). Psychological and cortisol responses to and recovery from exposure to a body image threat. SAGE Open. https://doi.org/10.1177/2158244016642378
- [Background] Marschall, D. E., Sanftner, J. L., & Tangney, J. P. (1994). The State Shame and Guilt Scale (SSGS). Fairfax, VA: George Mason University.
- [Background] Pearl RL, Puhl RM. Measuring internalized weight attitudes across body weight categories: validation of the modified weight bias internalization scale. Body Image. 2014 Jan;11(1):89-92. doi: 10.1016/j.bodyim.2013.09.005. Epub 2013 Oct 4. PMID 24100004
- [Background] Shaffer F, Ginsberg JP. An Overview of Heart Rate Variability Metrics and Norms. Front Public Health. 2017 Sep 28;5:258. doi: 10.3389/fpubh.2017.00258. eCollection 2017. PMID 29034226
- [Background] Wolpe, J., 1990. The Practice of Behavior Therapy, Rev. ed. Pergamon Press, New York.